CLINICAL TRIAL: NCT02356185
Title: Prevalence, Socio-demographic Correlates of Substance Use Disorders Among HIV-infected Adults in Cameroon, and Their Influence on Adherence to Antiretroviral Therapy and Immunological Feature: Study Protocol for a Retrospective Cohort Study
Brief Title: Substance Use Disorders in HIV People of Cameroon
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Goulfey Health District Unit (Other)
Collaborators: Yaounde Central Hospital (Other Government); Edea Regional Hospital (Other); University of Yaounde 1 (Other); NYU Langone Health (Other)
Responsible Party: Principal Investigator, Jean Joel R. Bigna, Head Officer, Goulfey Health District Unit
Other Study IDs: ASSIST-HIV
Record Dates: First submitted 2014-12-24; First posted 2015-02-05 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: HIV
Keywords: Alcohol Drinking; Injecting drug; Antiretroviral therapy; sub-Saharan Africa
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Background:

Data are scarce concerning injecting drug use (IDU) and alcohol consumption among HIV-infected people on highly active antiretroviral treatment (HAART) in Cameroon. The aim of this study is to determine the prevalence of alcohol consumption and IDU among HIV-infected people on HAART; to determine sociodemographic factors associated with alcohol abuse and IDU among people on HAART; and to determine impact of alcohol consumption and IDU on adherence to HAART.

Methods/Design:

The investigators will conduct a cross sectional study at the Yaoundé Central Hospital in Cameroon, from February to August 2015. Using a self-report questionnaire, the investigators will include at least 1,000 HIV-infected adults (18 years or more) on HAART for at least one month coming for HIV care. The investigators will exclude pregnant women. Data collection will include sociodemographic and economic profile, alcohol consumption using Alcohol Use Disorders Identification Test, injecting drug use, adherence to HAART using visual analog scale and self-rate report. The investigators will perform sub-analysis for sex group and area of habitation. A p value < 0.05 will be considered statistically significant.

Discussion:

There is a critical need of accurate estimates of the amplitude and the distribution of IDU and alcohol consumption among HIV-infected adults, in order to inform health policies maker for curbing burden of both injecting drug use and alcohol consumption among people living with HIV.

DETAILED DESCRIPTION:
1. Introduction

   1.1. Background

   In low and middle income countries, 28.6 million people were eligible for antiretroviral therapy (ART) based on 2013 guidelines and only around 10 million were currently on ART. Cameroon is a lower-middle-income country with a prevalence of human immunodeficiency virus (HIV) infection in adults of 4.3% in 2011. In the same year, coverage for antiretroviral therapy in adults and children was 49.6%, demonstrating the immensity of the work to be done to achieve the goals of good ART coverage. The considerable expansion of access to HIV treatment in the world has changed the epidemic of HIV infection. The importance of ART is well established. Life expectancy of adults receiving ART is approximately 80% of the normal life expectancy. The preventive effect of ART is increasingly evident, even in cases where the HIV epidemic is concentrated.

   There exists the link between alcohol consumption and infectious diseases, with the deleterious effect of alcohol on disease progression. In Cameroon, in general population, adult (15+ years) per capita alcohol consumption was 13.74 litters of pure alcohol. Heavy episodic drinking is 8.4% and 2.1% respectively among males and females in Cameroon in general population. Alcohol binge drinking was found in 11.6% of people living with HIV on ART and in 20.6% of those who were interrupted their treatment. Binge drinking was defined for male as consumption of 5 or more drinks, for female as consumption of 4 or more drinks, in about 2 hours. Alcohol use disorders screened with cutting down, annoyance by criticism, guilty feelings, eye-openers (cage) questionnaire are present among 17% of adults HIV-infected in Cameroon.

   In Cameroon, the prevalence of non-adherence to ART was 22.5% based on the Community Programs for Clinical Research on AIDS index and 34.9% based on the Centre for Adherence Support Evaluation index. Alcohol is one of the main factors of ART interruption and ART non-adherence. The consumption of alcohol being on ART decrease response to highly active ART, and decrease health related quality of life.

   In general, health data, including HIV prevalence data, are less robust for key populations than for general populations due to complexities in sampling (and lack of size estimation data), legal concerns and issues of stigma and discrimination. To date, studies on injecting drug user in Cameroon, and even in sub-Sahara Africa are scarce among HIV-infected people. The estimation showed that in 2012 worldwide about 12.7 million people had recently injected drugs and that, of these, 13.1% was living with HIV.

   1.2. Study rationale

   With this demonstrated burden so harmful of alcohol consumption and injecting drug use (IDU) among people living with HIV, it is necessary to measure the weight of alcohol consumption and IDU among HIV-infected adult on HAART; to understand why HIV-infected people consume alcohol and use injecting drug being on HAART in Cameroon, sub-Saharan Africa country; and to assess the impact of alcohol consumption and IDU on adherence to ART.
2. Study objectives

   The aim of this study is (1) to determine and describe the prevalence of alcohol consumption and IDU among HIV-infected people on HAART; (2) to determine sociodemographic factors associated with alcohol consumption and IDU among people on HAART; (3) and to determine impact of alcohol consumption and IDU on adherence to HAART.
3. Methods

   3.1. Design

   The investigators will use cross-sectional design. The recruitment of participants will be conducted from January to June 2015. Socio-demographic data, adherence to ART, alcohol consumption will be self-reported by the patients with a questionnaire, but patient will can ask more clarifications if he/she not understood a question. The investigators will follow STROBE guidelines for the report this study.

   3.2. Setting

   Cameroon is a sub-Saharan central Africa country, divided in ten region and with a population of 19,406,100 inhabitants in 2011. The adult prevalence rate of HIV in the country is 4.3%. In Yaoundé, capital of Cameroon, site of recruitment, the adult prevalence rate of HIV infection is 6.4% (3.6% for men and 8.9% for women). Subjects were recruited at Day Hospital in Yaoundé Central Hospital. It is the largest HIV clinic in the country. This is an urban center in the heart of Yaoundé city.

   3.3. Participants

   The investigators will include in this study subjects who are aged 18 years or above and who were on HAART for at least one month. The investigators will exclude pregnant women. Informed consent will be a prerequisite for participating in the study, and will be provided verbally.

   3.4. Data collection

   3.4.1. Sociodemographic profile

   The investigators will collect age, gender, sexual orientation, last level of education, monthly household income, area of habitation, number or person in household, mode of healthcare payment, marital status, employment status, probable route of HIV infection and when, and disclosure of HIV status.

   3.4.2. Alcohol consumption

   The investigators will use the Alcohol Use Disorders Identification Test (AUDIT) to identify subjects with at-risk, hazardous, or harmful drinking. AUDIT has a possible range from 0 to 40. A score ≤ 7 is classified as no current problem (low risk drinking), a score range between 8 - 15 is classified as probable current problem drinking (risky or hazardous drinking), a score range between 16 - 19 is classified as high risk or harmful drinking, and a score ≥ 20 as define harm and likely to be alcohol dependent. The investigators prefer to use self-reported questionnaire vs. interview questionnaire because it may produce more accurate answers, but patients who will not well understand a question, could ask more clarifications. The investigators will therefore use AUDIT screening instrument test to classify current drinkers as problem or non-problem drinkers at cut-off ≥ 8. Sensitivity and specificity of AUDIT is respectively 51%-97% and 78%-96%. The investigators will define as current drinkers, all patients who had consumed alcohol in the last 12 months.

   3.4.3. Adherence to antiretroviral therapy

   The investigators will use several methods to measure adherence to ART: a linear visual analogue scale (VAS) on the past month and self-rate of adherence to ART in the last month using scale from '1 - very good' to '5 - very bad'.

   3.4.4. Injecting drug use

   Patients will report if Yes or No, they have already used an injectable drug. If yes, they will give frequency and last time of use.

   3.5. Statistical analysis

   3.5.1. Sample size

   The sample calculation was based on alcohol consumption, because there is no data for IDU in Cameroon among HIV-infected people. The investigators assume that alcohol abuse among adults HIV-infected is 17%. With a 95% confidence interval (95%CI), acceptable difference of 5%; the minimal required sample size was 217 adult HIV-infected on ART. The investigators have used Windows Program for Epidemiologist (WinPepi, version 11.43) to estimate required sample size. Because the investigators will use self-reported questionnaire, the investigators suppose 20% for missing data. Therefore, the minimal required sample size will 272 for male and 272 for female because alcohol consumption was different between both sex (14). The investigators hope to have a sample of about 1,000 patients to have a high powered study.

   3.5.2. Statistical method

   Data will be coded, entered, and analyzed using the Statistical Package for Social Science version 20.0 for Windows (IBM Corp. Released 2011. IBM SPSS Statistics for Windows, Version 20.0. Armonk, New York: IBM Corp.). The investigators will describe continuous variables using means with standard deviations or using median with interquartile range, and categorical variables using their frequencies and percentages. For all tests, we will use 2-sided p-values with alpha < 0.05 level of significance. The investigators used χ² test or equivalents for categorical variables, Student T test for means, and Mann-Whitney U test for medians. Null hypothesis of no difference was rejected if the 95% CI of odds ratio (OR) estimates excluded 1. All regression analyses will be conducted with stepwise forward method with entry in model if p value ≤ 0.2. Multiple imputation will be used to handle missing data, creating a new data set which was the average of five data sets of imputed values. The investigators will only impute socio-demographic data for regression analysis.
4. Ethical considerations

   The study will be conducted in accordance with Helsinki Declaration. Prior to enrolment, all eligible participants will provide verbal consent. Patients with alcohol consumption, injecting drug use and/or non-adherence to ART will receive a counseling to address this problem according WHO recommendations.
5. Discussion

The expansion of the use of ART helped make HIV infection as a chronic disease. One of the major challenges to overcome is the effective use of ARVs to improve the outcome of people living with HIV. Consumption of alcohol and injecting drug by patients on HAART may be obstacles. The scientific evidence is already done for the first for its negative effect on antiretroviral therapy in others people than Africa but very few studies on the IDU are done, particularly in Africa. Even if there are data on alcohol consumption being on antiretroviral therapy exist in Africa, very few studies have a large sample size. More and to the best of our best knowledge, there are almost no studies on the prevalence of injecting drug use among HIV infected people in Africa, particularly in Cameroon.

With this study, the gap in knowledge about injecting drugs and alcohol and their effects on adherence to antiretroviral therapy may be addressed. This will guide future research. This knowledge can also provide to clinicians and policy makers of health, a light on the implementation of guidelines to improve the outcomes of people living with HIV in our context.

One of the limitations that might emerge during the implementation of this study is the presence of missing data, particularly related to data collection of the study by patients themselves. It is nonetheless necessary to use this form of data collection, since we will collect data on adherence to ARV treatment, on alcohol consumption, and on injecting drug use. In general, people tend to underestimate their alcohol consumption and overestimate adherence to treatment when a third party ask them a question about. In addition, the use of drugs is prohibited by law. Some patients may therefore deny its consumption. This is why no name or contact will be asked, no signature or written consent for participation in the study will be required for this study. We will thus use verbal consent.

The final report of this study in the form of scientific paper will be published in peer-reviewed journals. Findings will further be presented at conferences and submitted to relevant health authorities.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or older
* being for at least one month on highly active antiretroviral therapy

Exclusion Criteria:

* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected people
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Adherence to antiretroviral therapy | All days up to 180 days
  The investigators will measure adherence to antiretroviral therapy using a linear visual analogue scale on the past month as primary method of measure

SECONDARY OUTCOMES:
Self-rate of adherence to antiretroviral therapy | All days up to 180 days
  The investigators will measure adherence to antiretroviral therapy using self-rate by following scale: '1 - very good' to '5 - very bad'

OTHER OUTCOMES:
Alcohol consumption | All days up to 180 days
  The investigators will use the Alcohol Use Disorders Identification Test (AUDIT) to identify subjects with at-risk, hazardous, or harmful drinking. AUDIT has a possible range from 0 to 40. A score ≤ 7 is classified as no current problem (low risk drinking), a score range between 8 - 15 is classified as probable current problem drinking (risky or hazardous drinking), a score range between 16 - 19 is classified as high risk or harmful drinking, and a score ≥ 20 as define harm and likely to be alcohol dependent. The investigators prefer to use self-reported questionnaire vs. interview questionnaire because it may produce more accurate answers, but patients who will not well understand a question, could ask more clarifications. The investigators will therefore use AUDIT screening instrument test to classify current drinkers as problem or non-problem drinkers at cut-off ≥ 8.
Injecting drug use | All days up to 180 days
  Patients will report if Yes or No, they have already used an injectable drug. If yes, they will give frequency and last time of use.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Joel R Bigna, MD, Principal Investigator — Goulfey Health District Unit

REFERENCES:
- [Background] Johnson LF, Mossong J, Dorrington RE, Schomaker M, Hoffmann CJ, Keiser O, Fox MP, Wood R, Prozesky H, Giddy J, Garone DB, Cornell M, Egger M, Boulle A; International Epidemiologic Databases to Evaluate AIDS Southern Africa Collaboration. Life expectancies of South African adults starting antiretroviral treatment: collaborative analysis of cohort studies. PLoS Med. 2013;10(4):e1001418. doi: 10.1371/journal.pmed.1001418. Epub 2013 Apr 9. PMID 23585736
- [Background] Wood E, Braitstein P, Montaner JS, Schechter MT, Tyndall MW, O'Shaughnessy MV, Hogg RS. Extent to which low-level use of antiretroviral treatment could curb the AIDS epidemic in sub-Saharan Africa. Lancet. 2000 Jun 17;355(9221):2095-100. doi: 10.1016/S0140-6736(00)02375-8. PMID 10902622
- [Background] Donnell D, Baeten JM, Kiarie J, Thomas KK, Stevens W, Cohen CR, McIntyre J, Lingappa JR, Celum C; Partners in Prevention HSV/HIV Transmission Study Team. Heterosexual HIV-1 transmission after initiation of antiretroviral therapy: a prospective cohort analysis. Lancet. 2010 Jun 12;375(9731):2092-8. doi: 10.1016/S0140-6736(10)60705-2. Epub 2010 May 26. PMID 20537376
- [Background] Granich RM, Gilks CF, Dye C, De Cock KM, Williams BG. Universal voluntary HIV testing with immediate antiretroviral therapy as a strategy for elimination of HIV transmission: a mathematical model. Lancet. 2009 Jan 3;373(9657):48-57. doi: 10.1016/S0140-6736(08)61697-9. Epub 2008 Nov 27. PMID 19038438
- [Background] Cohen MS, Chen YQ, McCauley M, Gamble T, Hosseinipour MC, Kumarasamy N, Hakim JG, Kumwenda J, Grinsztejn B, Pilotto JH, Godbole SV, Mehendale S, Chariyalertsak S, Santos BR, Mayer KH, Hoffman IF, Eshleman SH, Piwowar-Manning E, Wang L, Makhema J, Mills LA, de Bruyn G, Sanne I, Eron J, Gallant J, Havlir D, Swindells S, Ribaudo H, Elharrar V, Burns D, Taha TE, Nielsen-Saines K, Celentano D, Essex M, Fleming TR; HPTN 052 Study Team. Prevention of HIV-1 infection with early antiretroviral therapy. N Engl J Med. 2011 Aug 11;365(6):493-505. doi: 10.1056/NEJMoa1105243. Epub 2011 Jul 18. PMID 21767103
- [Background] Kato M, Granich R, Bui DD, Tran HV, Nadol P, Jacka D, Sabin K, Suthar AB, Mesquita F, Lo YR, Williams B. The potential impact of expanding antiretroviral therapy and combination prevention in Vietnam: towards elimination of HIV transmission. J Acquir Immune Defic Syndr. 2013 Aug 15;63(5):e142-9. doi: 10.1097/QAI.0b013e31829b535b. PMID 23714739
- [Background] Rehm J, Parry CD. Alcohol consumption and infectious diseases in South Africa. Lancet. 2009 Dec 19;374(9707):2053. doi: 10.1016/S0140-6736(09)62150-4. No abstract available. PMID 20109832
- [Background] Samet JH, Walley AY, Bridden C. Illicit drugs, alcohol, and addiction in human immunodeficiency virus. Panminerva Med. 2007 Jun;49(2):67-77. PMID 17625483
- [Background] Samet JH, Horton NJ, Traphagen ET, Lyon SM, Freedberg KA. Alcohol consumption and HIV disease progression: are they related? Alcohol Clin Exp Res. 2003 May;27(5):862-7. doi: 10.1097/01.ALC.0000065438.80967.56. PMID 12766632
- [Background] Marcellin F, Boyer S, Protopopescu C, Dia A, Ongolo-Zogo P, Koulla-Shiro S, Abega SC, Abe C, Moatti JP, Spire B, Carrieri MP; EVAL Study Group. Determinants of unplanned antiretroviral treatment interruptions among people living with HIV in Yaounde, Cameroon (EVAL survey, ANRS 12-116). Trop Med Int Health. 2008 Dec;13(12):1470-8. doi: 10.1111/j.1365-3156.2008.02170.x. Epub 2008 Nov 5. PMID 19000156
- [Background] L'akoa RM, Noubiap JJ, Fang Y, Ntone FE, Kuaban C. Prevalence and correlates of depressive symptoms in HIV-positive patients: a cross-sectional study among newly diagnosed patients in Yaounde, Cameroon. BMC Psychiatry. 2013 Sep 22;13:228. doi: 10.1186/1471-244X-13-228. PMID 24053612
- [Background] Pefura-Yone EW, Soh E, Kengne AP, Balkissou AD, Kuaban C. Non-adherence to antiretroviral therapy in Yaounde: prevalence, determinants and the concordance of two screening criteria. J Infect Public Health. 2013 Aug;6(4):307-15. doi: 10.1016/j.jiph.2013.02.003. Epub 2013 Apr 22. PMID 23806707
- [Background] Azar MM, Springer SA, Meyer JP, Altice FL. A systematic review of the impact of alcohol use disorders on HIV treatment outcomes, adherence to antiretroviral therapy and health care utilization. Drug Alcohol Depend. 2010 Dec 1;112(3):178-93. doi: 10.1016/j.drugalcdep.2010.06.014. Epub 2010 Aug 11. PMID 20705402
- [Background] Hendershot CS, Stoner SA, Pantalone DW, Simoni JM. Alcohol use and antiretroviral adherence: review and meta-analysis. J Acquir Immune Defic Syndr. 2009 Oct 1;52(2):180-202. doi: 10.1097/QAI.0b013e3181b18b6e. PMID 19668086
- [Background] Neuman MG, Schneider M, Nanau RM, Parry C. Alcohol Consumption, Progression of Disease and Other Comorbidities, and Responses to Antiretroviral Medication in People Living with HIV. AIDS Res Treat. 2012;2012:751827. doi: 10.1155/2012/751827. Epub 2012 Mar 11. PMID 22496971
- [Background] Cook RL, Sereika SM, Hunt SC, Woodward WC, Erlen JA, Conigliaro J. Problem drinking and medication adherence among persons with HIV infection. J Gen Intern Med. 2001 Feb;16(2):83-8. doi: 10.1111/j.1525-1497.2001.00122.x. PMID 11251758
- [Background] Tran BX, Nguyen LT, Do CD, Nguyen QL, Maher RM. Associations between alcohol use disorders and adherence to antiretroviral treatment and quality of life amongst people living with HIV/AIDS. BMC Public Health. 2014 Jan 10;14:27. doi: 10.1186/1471-2458-14-27. PMID 24411007
- [Background] Samet JH, Horton NJ, Meli S, Freedberg KA, Palepu A. Alcohol consumption and antiretroviral adherence among HIV-infected persons with alcohol problems. Alcohol Clin Exp Res. 2004 Apr;28(4):572-7. doi: 10.1097/01.alc.0000122103.74491.78. PMID 15100608
- [Background] Kumar S, Jin M, Ande A, Sinha N, Silverstein PS, Kumar A. Alcohol consumption effect on antiretroviral therapy and HIV-1 pathogenesis: role of cytochrome P450 isozymes. Expert Opin Drug Metab Toxicol. 2012 Nov;8(11):1363-75. doi: 10.1517/17425255.2012.714366. Epub 2012 Aug 8. PMID 22871069
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. Bull World Health Organ. 2007 Nov;85(11):867-72. doi: 10.2471/blt.07.045120. PMID 18038077
- [Background] Fiellin DA, Reid MC, O'Connor PG. Screening for alcohol problems in primary care: a systematic review. Arch Intern Med. 2000 Jul 10;160(13):1977-89. doi: 10.1001/archinte.160.13.1977. PMID 10888972
- [Background] Cheng DM, Libman H, Bridden C, Saitz R, Samet JH. Alcohol consumption and lipodystrophy in HIV-infected adults with alcohol problems. Alcohol. 2009 Feb;43(1):65-71. doi: 10.1016/j.alcohol.2008.09.004. PMID 19185212
- See also: The World Bank. Cameroon data: The World Bank — http://data.worldbank.org/country/cameroon
- See also: WHO, UNICEF, UNAIDS. Global update on HIV treatment 2013: Results, impact and opportunities 2013 — http://www.who.int/iris/bitstream/10665/85328/1/WHO_HIV_2013.9_fre.pdf
- See also: National Institute of Alcohol Abuse and Alcoholism. NIAAA council approves definition of binge drinking: National Institute of Alcohol Abuse and Alcoholism; 2004 — http://pubs.niaaa.nih.gov/publications/Newsletter/winter2004/Newsletter_Number3.pdf
- See also: Babor TF, Higgins-Biddle JC, Saunders JB, Monteiro MG. AUDIT: The Alcohol Use Disorders Identification Test, Guidelines for Use in Primary Care. Geneva, Switzerland: World Health Organization; 2001 — http://whqlibdoc.who.int/hq/2001/who_msd_msb_01.6a.pdf